CLINICAL TRIAL: NCT06433349
Title: A Multi-center Investigation of Family Health, Needs, Perceived Support, Self-efficacy and Quality of Life During the Cancer Trajectory: A Longitudinal Mixed Methods Study Among Danish Cancer Patients and Their Caregivers
Brief Title: A Multi-center Investigation of Family Health.
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Sygehus Lillebaelt (Other); Zealand University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Laerke Kjaer Tolstrup, Principal investigator, Odense University Hospital
Other Study IDs: FaCe Cancer
Record Dates: First submitted 2024-02-23; First posted 2024-05-29 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Prostate Cancer; Colorectal Cancer; Hematologic Neoplasms; Caregivers
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Hematologic Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with breast-, prostate- colorectal cancer or lymphoma: Patients will complete the following questionnaires at baseline, 3, 6, 12, and 18 months:
  Family Health Scale (Long-form), the ICE Family Perceived Support Questionnaires, EQ-5D-5L, The general self-efficacy scale (GSE), the Patient Health Questionnaire-9 (PHQ-9), the National Comprehensive Cancer Network Distress thermometer (NCCN DT) and resilience was assessed with the Danish version of the 2-item Connor-Davidson-Resilience Scale (CD-RISC2).
  A subset of the patients will also participate in family interviews (n=12-15).
  Interventions: Other: Survey and interviews
- Caregivers to patients with breast-, prostate- colorectal cancer or lymphoma.: Caregivers will complete the following questionnaires at baseline, 3, 6, 12, and 18 months:
  Family Health Scale (Long-form), the ICE Family Perceived Support Questionnaires, EQ-5D-5L, The general self-efficacy scale (GSE), the Patient Health Questionnaire-9 (PHQ-9), the National Comprehensive Cancer Network Distress thermometer (NCCN DT) and resilience was assessed with the Danish version of the 2-item Connor-Davidson-Resilience Scale (CD-RISC2).
  A subset of the caregivers will also participate in family interviews (n=12-15).
  Interventions: Other: Survey and interviews

INTERVENTIONS:
Other: Survey and interviews — Questionnaires and interviews

SUMMARY:
The current healthcare system is unable to identify burdened and vulnerable families affected by cancer, partly due to a lack of knowledge of how cancer affects family health during treatment and survivorship. Recent reviews have documented a general lack of cancer studies including both the patient and the family, and a particular deficiency in studies including more than the spouse.

The principal aim of this study is to investigate family health, needs and perceived support, quality of life, self-efficacy, depression, stress and resilience in both patients with cancer and their families across the cancer trajectory. Additionally, the study seeks to identify particularly burdened and vulnerable families and investigate contributing factors to their vulnerability.

DETAILED DESCRIPTION:
Background Around 45,000 Danes are diagnosed with cancer each year with an increasing incidence and more than 350,000 people are living with cancer. Depending on the specific diagnosis, the 5-year survival rates range between 67% for men and 69% for women. Approximately 15,000 die of cancer each year.

Receiving a cancer diagnosis not only affects patients; it also affects family members, making cancer disorders a family affair. However, adult cancer research rarely focuses on the well-being and health of the whole family, which is worrying as one-third of the Danish population gets a cancer diagnosis before the age of 75, suggesting that most Danes will become caregivers to a cancer patient at some time during their lives. Adding to this, the Danish Cancer Society recently documented that patients who receive support from caregivers perform better on all parameters, i.e. patients are more aware of signs of relapse and get more frequent help when needed. Thus, caregiver support is a significant component for getting well through the course of cancer without unnecessary discomfort.

In addition, there is an increasing political focus on the efficient utilization of resources, which has resulted in fast-track treatments (Danish: Kræftpakker) and an increasing number of patients in outpatient clinics. This change of treatment setting from hospital to outpatient settings or even hospitalization in the homes of patients directly involves family caregivers in the care of the individual patient, i.e. with treatment, physical care, or emotional support. Thus, the future healthcare system will increasingly depend on the patient´s family and social network when supporting patients with cancer, ensuring, and supporting the health of individuals and communities in multiple inter-connected ways. This evident shift in responsibility from the public to the private sphere has a direct and substantial effect on family function, with a greater burden on the family members involved, which may eventually lead to deteriorated overall family health. Adding to this, there is growing evidence that the health and well-being of family caregivers are affected by higher expectations of active involvement in the care of their ill family member. Families confronted with health problems are at risk of stress and disturbance of family functioning that could cause other health problems and additional harm within the family system. Similarly and highly concerning, is evidence suggesting caregivers have high rates (42%) of depression, a disorder that in itself is associated with multiple concerning outcomes including premature death, chronic disease courses, self-harm, and suicides.

The current healthcare system is unable to identify burdened and vulnerable families affected by cancer, partly due to a lack of knowledge of how cancer affects family health during treatment and survivorship. Recent reviews have documented a general lack of cancer studies including both the patient and the family, and a particular deficiency in studies including more than the spouse.

The principal aim of this study is to investigate family health, needs and perceived support, quality of life, self-efficacy, depression, stress and resilience in both patients with cancer and their families across the cancer trajectory. Additionally, the study seeks to identify particularly burdened and vulnerable families and investigate contributing factors to their vulnerability.

Methods and material

Setting The study will recruit patients and caregivers from six different Danish hospital departments.

Participants In total, 240 patients and their appointed caregivers will be included. Inclusion criteria: curative intended patients and their eventual appointed caregivers >18 years affected by breast-, prostate-, colorectal cancer or lymphoma.

Exclusion criteria: Not able to understand or give written informed consent.

Design The Face Cancer study is a multi-center investigation of family health, needs, perceived support, self-efficacy, stress, resilience, and quality of life during the cancer trajectory among Danish cancer patients and their adult family caregivers. The study will use mixed methods including patient-reported outcomes in a longitudinal, prospective multicenter survey combined with family interviews conducted in a subset of participants included in the survey. A sequential explanatory design will be applied involving two phases, wherein the quantitative data collection (survey) and analysis will be followed by qualitative follow-up (interviews). Thus, the qualitative data from the family interviews will help to explain and interpret the context and depth of the mechanisms underlying the survey results. The rationale for applying a mixed-methods approach is to gain a deeper and more comprehensive understanding of the impact of cancer on patients and their families. For data presentation purposes, it will be depicted, by the use of a joint display, how the quantitative data is used to inform the qualitative data collection.

Quantitative data A prospective longitudinal multicenter survey including curatively intended cancer patients from the target group and their appointed adult family member(s) at entry of treatment (baseline), during treatment (3 months), and at 6, 12, and 18 months after baseline. The survey includes the following questionnaires. Family-reported outcomes will be assessed by the translated and validated Family Health Scale (Long-form) including family social and emotional health processes, family healthy lifestyle, family health resources, and family external social supports. Perceived support will be assessed by the ICE Family Perceived Support Questionnaires. HRQoL is assessed by the short generic EQ-5D-5L (EuroQol-5 dimensions). Self-efficacy is measured by the Danish version of the ten-item validated general self-efficacy scale (GSE) questionnaire to investigate the ability to act towards problems in everyday life. The GSE covers a broad range of the sense of personal competence to deal effectively with stressful situations. The scale has been found to have high validity and reliability in various populations across contexts and cultures To assess the degree of depression, the Patient Health Questionnaire-9 (PHQ-9) will be used. The Level of distress was measured with the Danish version of the National Comprehensive Cancer Network Distress thermometer (NCCN DT), and resilience was assessed with the Danish version of the 2-item Connor-Davidson-Resilience Scale (CD-RISC2). The survey will also assess real-time family needs & preferences in free text.

In total, 240 patients (60 patients per patient group) plus appointed family members will be included based on a power calculation of SD applied sqrt(2)*22 = 31 in the Family Health Scale. This would require 44 patients per patient group plus dropouts with 90% power to detect a minimal clinically important difference change two-time any pair of two-time points in the longitudinal design. Data are collected from six confirmed sites (Danish cancer departments) and questionnaires are distributed via the national mailbox e-Boks.

Qualitative data Family interviews will be conducted to illuminate how patients and caregivers experience (perceive) vulnerable situations, their family supportive care needs, and family support during and after cancer treatment. The groups (n=12-15) will consist of families (one patient and either one or two caregivers) identified in the survey. The interviews will take place longitudinally at two time points at three months (during treatment) and 12 months (during follow-up) after the completion of baseline questionnaires. The interviews can take place either at the hospital, in the patients´ homes or online depending on the preferences of patients and relatives, and are expected to last approximately one hour. We plan to use an integrated approach combining phenomenology with hermeneutics to gain a more complete understanding of the families' experiences, recognizing both their subjective perceptions and the broader cultural and social significance. We will try to carry out the interviews inductively, letting the respondents reflect on their own experiences without imposing preconceived notions. An interview guide will be prepared in alignment with this and the family systems theory. Purposive sampling will be used to ensure the inclusion of families with maximal variation in age, gender, and family life situation will be invited. Thematic analysis by Braun and Clarke is chosen to extract data, identify patterns, and analyze data and themes. NVivo will be used for coding interview data.

ELIGIBILITY:
Inclusion Criteria:

* curative intended patients and their eventual appointed caregivers >18
* breast-, prostate- colorectal cancer or lymphoma.

Exclusion Criteria:

* Not able to understand or give written informed consent
* Not able to speak Danish or complete questionnaires in Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast, prostate, colorectal cancer, or lymphoma and their appointed caregivers. The patients are to receive anti-neoplastic treatment with curative intent at one of the six hospitals included sites.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To investigate family health during the cancer trajectory. | 1 year
  The Family Health Scale: For each dimension, sum the scores to get a total score. Higher scores indicate better health. The ICE Family Perceived Support Questionnaires: Sum the scores for each item to get a total score. Higher scores indicate higher perceived support. The EQ-5D-5L: Digits for the five dimensions can be combined into a number that describes the patient's health from 11111 (full health) to 55555 (worst health). The General self-efficacy scale: Ranges between 10 and 40, a higher score indicating more self-efficacy. The Patient Health Questionnaire-9: Score ranges from 0 to 27 (5-9 are mild depression; 10-14 as moderate; 15-19 as moderately severe; ≥ 20 as severe). The National Comprehensive Cancer Network Distress thermometer, a single-item tool using a 0 (no distress) to 10 (extreme distress). The 2-item Connor-Davidson-Resilience Scale: Each item has a score between 0 and 4. Total scores are calculated by the two items. A higher score indicates higher resilience.

SECONDARY OUTCOMES:
to identify vulnerable families and examine determinants for their vulnerability at identifying vulnerable families. To identify vulnerable families | 1 year
  To identify vulnerable families for the interviews, data from the survey will be used in accordance with the explanatory sequential design. To identify vulnerable patients and caregivers from the PRO-results, 10 items from the Family Health Scale long-form (items 4, 11, 16, 17, 18, 23, 26, 27, 31, 32), which corresponds to the Family Health short form, will be used. Each participant can have a final family health score between 0 and 10 points. Poor family health = 0-5 points; moderate family health = 6-8 points; excellent family health = 9-10 points [30]. If either the patient or the caregiver has a score indicating poor or moderate family health, the family will be considered a candidate for the interviews. Following this identification, interviews will be carried out to elucidate determinant factors for their vulnerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No
This project generates data from human subjects, including (e.g., interview transcripts and survey responses). These data contain sensitive and personally identifiable information.
  The data will not be shared publicly due to participant confidentiality.
  Standard institutional practices will be used for file naming, version control, and documentation. Metadata will be maintained internally for project management purposes but will not be shared externally.
  No public or external data sharing is planned. Data access will be limited to the study team, in compliance with approval of the Danish Data Protection Agency (23/52139). The and participant consent agreements.
  Data will be stored securely stored at a secure logged server at Open Patient data Explorative Network (OP_2013), Department of Clinical Research, University of Southern Denmark with access restricted to authorized project personnel.
  Data security and compliance will be overseen by the Principal Investigator in coordinat

REFERENCES:
- [Result] Coyne E, Heynsbergh N, Dieperink KB. Acknowledging cancer as a family disease: A systematic review of family care in the cancer setting. Eur J Oncol Nurs. 2020 Dec;49:101841. doi: 10.1016/j.ejon.2020.101841. Epub 2020 Oct 14. PMID 33130424
- [Result] Adashek JJ, Subbiah IM. Caring for the caregiver: a systematic review characterising the experience of caregivers of older adults with advanced cancers. ESMO Open. 2020 Sep;5(5):e000862. doi: 10.1136/esmoopen-2020-000862. PMID 32963088
- [Result] Weiss-Laxer NS, Crandall A, Okano L, Riley AW. Building a Foundation for Family Health Measurement in National Surveys: A Modified Delphi Expert Process. Matern Child Health J. 2020 Mar;24(3):259-266. doi: 10.1007/s10995-019-02870-w. PMID 31912378
- [Result] Jansen L, Dauphin S, van den Akker M, De Burghgraeve T, Schoenmakers B, Buntinx F. Prevalence and predictors of psychosocial problems in informal caregivers of older cancer survivors - A systematic review: Still major gaps in current research. Eur J Cancer Care (Engl). 2018 Nov;27(6):e12899. doi: 10.1111/ecc.12899. Epub 2018 Aug 31. PMID 30168877
- [Result] Gray TF, Azizoddin DR, Nersesian PV. Loneliness among cancer caregivers: A narrative review. Palliat Support Care. 2020 Jun;18(3):359-367. doi: 10.1017/S1478951519000804. PMID 31581964
- [Result] Ochoa CY, Buchanan Lunsford N, Lee Smith J. Impact of informal cancer caregiving across the cancer experience: A systematic literature review of quality of life. Palliat Support Care. 2020 Apr;18(2):220-240. doi: 10.1017/S1478951519000622. PMID 31588882
- [Result] Cochrane A, Reid O, Woods S, Gallagher P, Dunne S. Variables associated with distress amongst informal caregivers of people with lung cancer: A systematic review of the literature. Psychooncology. 2021 Aug;30(8):1246-1261. doi: 10.1002/pon.5694. Epub 2021 May 4. PMID 33945184
- [Result] Northouse L, Williams AL, Given B, McCorkle R. Psychosocial care for family caregivers of patients with cancer. J Clin Oncol. 2012 Apr 10;30(11):1227-34. doi: 10.1200/JCO.2011.39.5798. Epub 2012 Mar 12. PMID 22412124
- [Result] Geng HM, Chuang DM, Yang F, Yang Y, Liu WM, Liu LH, Tian HM. Prevalence and determinants of depression in caregivers of cancer patients: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Sep;97(39):e11863. doi: 10.1097/MD.0000000000011863. PMID 30278483
- [Result] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Result] Konradsen H, Brodsgaard A, Ostergaard B, Svavarsdottir E, Dieperink KB, Imhof L, Luttik ML, Mahrer-Imhof R, Garcia-Vivar C. Health practices in Europe towards families of older patients with cancer: a scoping review. Scand J Caring Sci. 2021 Jun;35(2):375-389. doi: 10.1111/scs.12855. Epub 2020 Apr 14. PMID 32291782
- [Derived] Tolstrup LK, Hyldig N, Moller S, Stie M, Kjerholt M, Jarden M, Piil K, Coyne E, Garcia-Vivar C, Voltelen B, Munk-Olsen T, Dieperink KB. Exploring family health, support, self-efficacy and quality of life during the cancer trajectory: a protocol for a longitudinal mixed methods multi-centre cohort study. BMJ Open. 2025 Oct 23;15(10):e102387. doi: 10.1136/bmjopen-2025-102387. PMID 41146379